CLINICAL TRIAL: NCT02024698
Title: Multi-center Clinical Evaluation of PC 1-Day vs 1-Day Acuvue Moist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-43
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- omafilcon A (Active Comparator): Study participants are randomized to wear omafilcon A lenses.
  Interventions: Device: omafilcon A
- etafilcon A (Active Comparator): Study participants are randomized to wear etafilcon A lenses.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: omafilcon A — contact lens
  Other Names: Proclear 1 Day (omafilcon A)
  Arms: omafilcon A
Device: etafilcon A — contact lens
  Other Names: 1-Day Acuvue Moist (etafilcon A)
  Arms: etafilcon A

SUMMARY:
The objective of this study is to compare the clinical performance of ProClear 1-Day versus 1-Day Acuvue Moist each for one week of daily disposable wear.

DETAILED DESCRIPTION:
The purpose of this cross-over study is to evaluate the clinical performance of the ProClear-1 Day in comparison with 1-Day Acuvue® Moist®. In particular, the study will focus on lens wearing comfort.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Have the use of a mobile phone to send and receive text messages throughout the day for the duration of the study.
* Has had a self-reported visual exam in the last two years
* Is an adapted soft CL (Contact Lens) wearer
* Must be able to wear their lenses at least 6 full days over the 7 days; 14 hours per day, assuming there are no contraindications for doing so
* Has a CL spherical prescription between - 1.00 and - 6.00 (inclusive)
* Has less than 0.75D (Diopters) spectacle cylinder in each eye.
* Is correctable to a visual acuity of 20/25 or better in both eyes
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Is willing to comply with the wear schedule (at least 40 hrs per week)
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a CL prescription outside the range of - 1.00 to -6.00D
* Has a spectacle cylinder greater than -0.50D of cylinder in either eye.
* Has best corrected spectacle distance vision worse then 20/25 in either eye.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars.
* Is aphakic.
* Is presbyopic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Siegel, OD, Principal Investigator — Sun City West Eye Care
Locations (4):
- United States (4):
  - Phoenix Eye Care, PLLC, Phoenix, Arizona
  - Lake Zurich Eye Care, Lake Zurich, Illinois
  - Drs. Quinn, Foster & Assoc., Athens, Ohio
  - Vision Professionals, New Albany, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Etafilcon A First, Then Omafilcon A: Study participants are randomized to wear etafilcon A pair of study lenses then crossover to the alternate pair.
- Omafilcon A First, Then Etafilcon A: Study participants are randomized to wear omafilcon A pair of study lenses then crossover to the alternate pair.
Period: First Intervention (7 Days)
Arm/Group | Etafilcon A First, Then Omafilcon A | Omafilcon A First, Then Etafilcon A
Started | 16 | 27
Completed | 16 | 26
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention (7 Days)
Arm/Group | Etafilcon A First, Then Omafilcon A | Omafilcon A First, Then Etafilcon A
Started | 16 | 26
Received Etafilcon A Twice | 1 | 0
Completed | 16 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Group: Study participants are randomized to wear omafilcon A or etafilcon A pair of study lenses then crossover to the alternate pair.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Comfort (Subjective Assessment)
Description: Subjective Assessment of comfort on insertion at baseline for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very uncomfortable, 10=cannot feel)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 42 | 43
units on a scale | 9.12 (1.17) | 9.16 (1.17)

2. Primary Outcome: Comfort (Subjective Assessment)
Description: Subjective Assessment: Insertion Comfort, Comfort During Day, Comfort Prior to Removal, Comfort Overall for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very uncomfortable, 10=cannot feel)
Time Frame: 1 Week
Population: One participant received etafilcon A twice which explains the uneven number of participants analyzed in the study results for week 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale
  Insertion Comfort | 9.15 (1.24) | 8.65 (1.77)
  Comfort During Day | 8.12 (2.00) | 8.63 (1.50)
  Comfort Prior to Removal | 7.20 (2.63) | 7.70 (1.95)
  Comfort Overall | 7.84 (1.75) | 8.28 (1.58)

3. Primary Outcome: Hydration (Subjective Assessment)
Description: Subjective Assessment of hydration on insertion at baseline for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very dehydrated, not hydrophilic, very dry, 10=very hydrated, ultra hydrophilic)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 42 | 43
units on a scale | 9.21 (1.02) | 9.35 (1.09)

4. Primary Outcome: Hydration (Subjective Assessment)
Description: Subjective Assessment: Initial Hydration, Hydration During Day, Hydration Prior to Removal for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very dehydrated, not hydrophilic, very dry, 10=very hydrated, ultra hydrophilic)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale
  Initial Hydration | 9.41 (1.00) | 8.84 (1.41)
  Hydration During Day | 8.02 (1.88) | 8.47 (1.37)
  Hydration Prior to Removal | 7.32 (2.44) | 7.53 (1.91)

5. Primary Outcome: Vision Quality (Subjective Assessment)
Description: Subjective Assessment: Visual quality on insertion at baseline for each pair using questionnaire and rated on subjective response scale (0-10; 0= clear vision, 10=perfectly sharp)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 42 | 43
units on a scale | 9.33 (1.59) | 9.16 (1.79)

6. Primary Outcome: Vision Satisfaction (Subjective Assessment)
Description: Subjective Assessment: Vision Satisfaction for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very unsatisfied, 10=very satisfied)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale | 9.07 (1.46) | 9.05 (1.34)

7. Primary Outcome: Dryness (Subjective Assessment)
Description: Subjective Assessment: Dryness During Day, Dryness Prior to Removal, Overall Dryness for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very dry, 10=no dryness)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale
  Dryness During Day | 8.05 (1.92) | 8.58 (1.48)
  Dryness Prior to Removal | 7.24 (2.43) | 7.70 (1.78)
  Overall Dryness | 7.71 (2.06) | 8.14 (1.71)

8. Primary Outcome: Handling (Subjective Assessment)
Description: Subjective Assessment: Handling on Insertion and Removal, Overall Handling for each pair using questionnaire and rated on subjective response scale. (0-10; 0= very difficult, 10=very easy)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale
  Insertion and Removal | 8.85 (1.99) | 8.44 (1.79)
  Overall | 8.85 (1.99) | 8.51 (1.75)

9. Primary Outcome: Eye Whiteness/Redness (Subjective Assessment)
Description: Subjective Assessment: Eye Whiteness/Redness for each pair using questionnaire and rated on subjective response scale. (0-10; 0= significant redness, 10=totally white)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
units on a scale | 8.63 (1.65) | 9.26 (1.11)

10. Primary Outcome: Overall Sensation of Smoothness (Subjective Assessment)
Description: Subjective Assessment: Overall sensation of smoothness at 1 week wear for each pair when asked "How would you rate the overall sensation of smoothness (deposit resistance) of the first study lenses, over the last week of wear?" (Likert 1-5; 1=excellent, 2=good, 3=average, 4=below average, 5=poor)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
participants
  Excellent | 25 | 24
  Good | 11 | 7
  Average | 2 | 9
  Below Average | 3 | 3
  Poor | 0 | 0

11. Primary Outcome: Overall Satisfaction for Lens
Description: Subjective Assessment: Satisfaction overall at 1 Week wear for each pair when asked "Overall, how satisfied was the subject with the study lenses, during the last week, with regards to: Overall?" (Likert 1-4; 1=completely satisfied, 2=somewhat satisfied, 3=somewhat dissatisfied, 4=completely dissatisfied)
Time Frame: 1 Week
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Omafilcon A | Etafilcon A
Number analyzed (Participants) | 41 | 43
participants
  Completely Satisfied | 17 | 21
  Somewhat Satisfied | 18 | 14
  Somewhat Dissatisfied | 5 | 7
  Completely Dissatisfied | 1 | 1

ADVERSE EVENTS:
Time Frame: From dispense up to one week for each study lenses
Arm/Group | Omafilcon A | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.